CLINICAL TRIAL: NCT00372814
Title: Adherence to IDDM Regimen in Urban Youth
Brief Title: Study of Intensive, Home-Based Family Therapy to Improve Illness Management in Youth With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deborah Ellis, Ph.D., Professor of Pediatrics, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DK59067B (completed); R01DK059067 (NIH)
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Insulin Dependent
Keywords: diabetes; regimen adherence; metabolic control; adolescents; family therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multisystemic Therapy (MST) (Experimental): Adolescents receiving MST will receive Intensive Home-Based Family Therapy which will consist of home-based, family psychotherapy sessions 2-3 times a week, lasting 60 minutes in duration from a pediatric mental health worker for six months. The purpose of the therapy sessions are to improve the youths' ability to complete their daily diabetes illness management tasks, reduce average blood glucose levels and improve metabolic control.
  Interventions: Behavioral: Intensive Home-Based Family Therapy
- Telephone Support Calls (Active Comparator): Adolescents receiving Supportive Telephone Calls (TS) will receive weekly 30 minute phone calls from a pediatric mental health worker for six months. The purpose of the call is to provide emotional support regarding the adolescent's chronic medical condition, assess adherence to the prescribed regimen and to help the adolescent brainstorm solutions to any barriers they identify to completion of diabetes care.
  Interventions: Behavioral: Supportive Telephone Calls

INTERVENTIONS:
Behavioral: Intensive Home-Based Family Therapy — Multisystemic Therapy (MST): Adolescents receiving MST will receive home-based, family psychotherapy sessions 2-3 times a week, lasting 60 minutes in duration from a pediatric mental health worker for six months. The purpose of the therapy sessions are to improve the youths' ability to complete their dilay diabetes illness management tasks, reduce average blood glucose levels and improve metabolic control.
  Other Names: Multisystemic Therapy, MST
  Arms: Multisystemic Therapy (MST)
Behavioral: Supportive Telephone Calls — Telephone Support Calls: Adolescents receiving TS will receive weekly 30 minute phone calls from a pediatric mental health worker for six months. The purpose of the call is to provide emotional support regarding the adolescent's chronic medical condition, assess adherence to the prescribed regimen and to help the adolescent brainstorm solutions to any barriers they identify to completion of diabetes care.
  Other Names: TS
  Arms: Telephone Support Calls

SUMMARY:
The study is a randomized clinical trial testing the effectiveness of Multisystemic Therapy (MST) for improving the treatment adherence, metabolic control and quality of life of urban adolescents with poorly controlled insulin dependent diabetes.

DETAILED DESCRIPTION:
The deterioration in regimen adherence and metabolic control associated with the adolescent developmental period is well-documented. However, a subset of high-risk adolescents with diabetes demonstrate much more serious adherence problems, as evidenced by chronically poor metabolic control (CPMC) and post-diagnostic admissions for diabetic ketoacidosis (DKA). Adolescents in CPMC represent a group at high risk for both short and long term diabetes complications and are therefore heavy users of medical resources and health care dollars. Minority and low-income children are over-represented among adolescents with CPMC.

The design for the proposed study is a randomized, controlled trial with a repeated measures design using a sample of 170 adolescents, 85 of whom will receive MST and 85 of whom will receive a telephone intervention to test the effect of increased attention (control condition). Subjects must have a current hemoglobin A1C (HbA1c) of >8% and an average HbA1c of >8% during the past year, must be diagnosed with insulin dependent diabetes for at least one year, be 10-17 years of age and reside in the metro Detroit tri-county area. Exclusion criteria are severe mental impairment/thought disorder, non-English speaking patient/parent or a co-morbid major medical condition such as cystic fibrosis. Families who are randomized to MST receive intensive, home-based family therapy for approximately six months. MST is a community based treatment originally designed for use with adolescents presenting with serious mental health problems, but which is adapted in the present study for use with chronically ill youth and serious adherence difficulties. Therapists meet with families two to three times per week at the beginning of treatment with a decreasing number of sessions at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* insulin dependent Type 1 or Type 2 diabetes
* diagnosed with diabetes ≥ 1 year
* current HbA1c ≥ 8%
* average HbA1c ≥ 8% over the past year
* aged 10 -17
* patient of Children's Hospital of Michigan Diabetes Clinic
* lives within 30 miles of Children's Hospital of Michigan

Exclusion Criteria:

* moderate to severe mental retardation (unable to complete study measures)
* psychosis or current suicidal intent
* any medical diagnosis that alters standard diabetes care

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2007-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Metabolic Control: Hemoglobin A1c (HbA1c) | treatment termination, 6-month follow up
  Retrospective measure of blood glucose control, encompasses the previous 2-3 months

SECONDARY OUTCOMES:
BMI percentile | treatment termination, 6-month follow up
  Body mass index (BMI) a value derived from the mass and height of an individual
Diabetes-Specific Family Functioning | treatment termination, 6-month follow up
  Diabetes Family Responsibility Questionnaire (DFRQ), Parental Monitoring of Adolescent Diabetes Care (PMADC), Diabetes Social Support Questionnaire-Family (DSSQ-Family)
DKA admissions and emergency room (ER) Visits: hospital information systems data extraction, Service Utilization Questionnaire (SUQ) | treatment termination, 6-month follow up
  The number of patient visits to acute care settings represents a significant health care cost in this high-risk population.
Regimen Adherence: Diabetes Management Scale (DMS), Twenty-Four Hour Recall Interview, Glucose Meter Downloads | treatment termination, 6-month follow up
  The DMS assesses a broad range of management behaviors, such as insulin management, dietary management, blood glucose monitoring, symptom response, and parent assistance/supervision. Glucose meters only assess blood glucose monitoring, but are empirically linked to metabolic control.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Ellis, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ellis DA, Naar-King S, Chen X, Moltz K, Cunningham PB, Idalski-Carcone A. Multisystemic therapy compared to telephone support for youth with poorly controlled diabetes: findings from a randomized controlled trial. Ann Behav Med. 2012 Oct;44(2):207-15. doi: 10.1007/s12160-012-9378-1. PMID 22644587
- [Result] Carcone AI, Ellis DA, Chen X, Naar S, Cunningham PB, Moltz K. Multisystemic Therapy Improves the Patient-Provider Relationship in Families of Adolescents with Poorly Controlled Insulin Dependent Diabetes. J Clin Psychol Med Settings. 2015 Sep;22(2-3):169-78. doi: 10.1007/s10880-015-9422-y. PMID 25940767